CLINICAL TRIAL: NCT01692080
Title: Implementation of an Asthma Program to Improve Asthma Identification and Education in Children
Status: Completed | Type: Observational
Sponsor: Duquesne University (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: DU Protocol #10-11
Record Dates: First submitted 2012-08-07; First posted 2012-09-25 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Asthma; Hypertension; Obesity
MeSH Terms: conditions — Asthma; Hypertension; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Asthma Screenings and Camps: Children, ages 5-17 years who participate in one of the asthma screenings or camps are eligible to participate in this study.
  Interventions: Behavioral: Asthma education

INTERVENTIONS:
Behavioral: Asthma education — Two separate asthma education classes are conducted to target two age groups: 6-10 yrs and 10-15 yrs. With the guidance of pharmacy faculty, student pharmacists develop innovative educational activities directed at three of the most common barriers to proper asthma control: avoidance of asthma triggers; compliance with asthma medications and proper usage of inhalers; and the importance of an asthma action plan. There is a different group of student pharmacists participating in each camp and this allows for variation in educational activities, all reinforcing the same important aspects of optimal asthma management. Students create age-appropriate activities for each group. Parents are required to attend camps with their child and participate in the asthma education sessions.
  Other Names: asthma knowledge intervention

SUMMARY:
The primary objective of this study is to document the prevalence and associations between asthma, hypertension, and obesity in children living in Pittsburgh, Pennsylvania and its surrounding regions.

The secondary objective is to determine the impact of various educational interventions on child and caregiver knowledge of asthma.

DETAILED DESCRIPTION:
The Asthma Program will consist of six screenings and three camps each year, for two consecutive years. Screenings will be conducted in areas where populations are known to be at increased risk for asthma and its complications, such as inner-city, lower socioeconomic, African-American populations. Screenings will be conducted at churches or schools in these areas one month prior to each camp in an effort to identify children with undiagnosed or uncontrolled asthma and refer them to the camps. Camps will also be conducted in areas where populations are known to be at increased risk for asthma and its complications to improve ease of access. Asthma and smoking cessation education will be provided at each camp to children and caregivers. Baseline data will be collected at each camp and assessed. Longitudinal clinical outcomes will be assessed in children attending multiple camps.

ELIGIBILITY:
Inclusion Criteria:

* Children, ages 5- 17 years attending the asthma camps and screenings.

Exclusion Criteria:

* Children younger than 5 years of age and adults 18 years of age and older.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Two screenings will be held prior to each camp, at two separate locations, for a total of six screenings per year. Screenings will be held at different locations throughout the city of Pittsburgh in an effort to increase identification and recruitment for subsequent camps. All children will be invited to participate in screenings, regardless of participation in the study. All children, ages 5-17 years, will be included in our study pending informed consent and assent. Camps will take place three times each year. All children will be invited to participate in camps, regardless of participation in the study. All children, ages 5-17 years will be included in our study pending informed consent and assent.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study is to document the prevalence of asthma, hypertension and obesity in children living in Pittsburgh's inner-city. | Up to three years

SECONDARY OUTCOMES:
The secondary outcome of this study is to determine the impact of various educational interventions on child and caregiver knowledge of asthma. | up to three years
  A pre and post asthma knowledge test will be given to children and caregivers prior to and after participation in the educational session conducted at each asthma camp. A paired sample t-test was used for comparison of pre and post knowledge tests and a p value of less than 0.05 will be considered to indicate a statistically significant difference.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer P Elliott, PharmD, Principal Investigator — Duquesne University
Locations (1):
- Duquesne University, Pittsburgh, Pennsylvania, United States